CLINICAL TRIAL: NCT05462847
Title: Comparing the Hemodynamic Effects of Volume Loading vs Non-loading During Induction of Anesthesia in Fluid Responder Patients With Coronary Artery Disease Undergoing Elective Coronary Artery Bypass Graft Surgery: a Randomized Controlled Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ayman Abougabal, Dr Abougabal, Kasr El Aini Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MS-618-2021
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Post Induction Hypotension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Volume loading (Experimental)
  Interventions: Drug: Ringer acetate
- Control (Active Comparator)
  Interventions: Drug: Ringer acetate

INTERVENTIONS:
Drug: Ringer acetate — 8ml/kg Ringer acetate over 10 minutes

SUMMARY:
All preoperative cardiac medications will be continued till the morning of the surgery, except angiotensin converting enzyme inhibitors. Patients will be pre-medicated with intramuscular morphine at 0.1 mg.kg-1 one hour before surgery. Upon arrival to the operating room, Initial monitoring included five lead electrocardiograms, non-invasive blood pressure, and pulse oximetry. At the attending anesthetists discretion, intravenous midazolam (0.05 mg/kg) will be administered for anxiolysis. Under local anesthesia an arterial line will be placed in the right radial artery and central venous line will be placed in the right internal jugular vein.

Before induction of anesthesia for all study patients, Electrical cardiometry device (ICON; Cardiotonic, Osypka; Berlin, Germany) will be applied to the patient through 4 electrodes at the following sites: Below the left ear, Above the midpoint of the left clavicle, Left mid-axillary line at level of the xiphoid process and 5 cm inferior to the third electrode. Stroke volume variability (SVV) was measured while patient maintaining standard calm breathing at 8 breath/minute for one-minute. Patients with SVV less than 13% will be excluded from the study. Thus, all patients included will be considered fluid responders[5]. The baseline data in the form of heart rate, systolic, diastolic, and mean systemic arterial pressures, CO, CI, SV, SVI, SVV, SVR, and SVRI will be recorded during the study period in all the patients.

Patients will then be randomly divided into two groups; control group will receive nothing before induction, while patients in volume loading group will receive volume loading of 8ml/kg Ringer acetate over 10 minutes. The volume loading will be repeated until SVV would be below 13%. The volume loading would be given by an anesthesia resident not involved in data collection.

For induction, Patients in both groups will receive 3 mcg/kg of fentanyl. Then in all patients, propofol will be injected slowly at 1.5 mg/kg in 0.25 mg/kg increments every 20 s till clinical loss of consciousness. Clinical loss of consciousness (defined as no response to auditory command) will be assessed by asking the patients repeatedly every 20 s to open their eyes. After loss of consciousness, atracurium 0.5 mg/kg will be administered to facilitate tracheal intubation. The stress response to laryngoscopy and tracheal intubation is secondary to marked increase in sympathetic activity and manifested in general as tachycardia and hypertension and will be managed with increments 0..25mcg fentanyl. Hemodynamic changes; 20 beats/ minute or 20 mmHg difference in heart rate and blood pressure respectively were considered to be significant. Anesthesia will be maintained by isoflurane (1-1.2 %). Patients will be mechanically ventilated to have target of PO2 above 300mmhg and PCO2 between 35-40mmg.

Any episode of hypotension (defined as mean arterial pressure [MAP] < 80% of the baseline reading and/or MAP <60 mmHg) will be managed by 5 mcg norepinephrine (which could be repeated if hypotension persists for 2 minutes).

If bradycardia occurred (defined as heart rate less than 50 bpm), it will be managed by IV atropine bolus (0.5 mg).

Hemodynamic data will be recorded 1-minte before the induction, 1-and 2-minutes after loss of consciousness, 1-minutes after intubation, then every 2-minutes for 15-minutes after intubation., the end point of the present study. Throughout this period the lungs will be mechanically ventilated with 50% air-oxygen mixture, to maintain an end-tidal carbon dioxide between 35 and 40 mmHg.

ELIGIBILITY:
Inclusion Criteria:

* patients with coronary artery disease ASA physical status III-IV scheduled for elective CABG surgery.

Exclusion Criteria:

* • left ventricular systolic dysfunction (LVSD) <40%,

  * persistent serious arrhythmias,
  * congestive cardiac failure, on mechanical ventilation,
  * intra-aortic balloon pump (IABP),
  * emergency surgery,
  * un controlled diabetes (HbA1C >8)
  * those with known allergy to any of the study's drugs,
  * severe systemic non-cardiac disease,

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Incidence of post-induction hypotension | 15 minutes
  Incidence of post-induction hypotension from start of induction of anesthesia till 15-minutes

SECONDARY OUTCOMES:
Incidence of post-induction hypertension, bradycardia, and tachycardia | 15 minutes
  Incidence of post-induction hypertension, bradycardia, and tachycardia

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Abougabal, Principal Investigator — lecturer of anesthesia Kasr Al Ainy hospital
Locations (1):
- Kasr Al Ainy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided